CLINICAL TRIAL: NCT06109246
Title: The Patient Enablement Instrument for Back Pain Turkish Version, Validity and Reliability Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_09
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most people experience low back pain at some point in their lives, and most low back pain is classified as nonspecific because the factor causing the pain cannot be identified. Current guidelines recommend self-management interventions for the management of nonspecific low back pain. The most commonly used assessment measures measure pain, disability, and quality of life. However, it is important to evaluate patients' ability to manage their nonspecific LBP-specific disease.

In 1997, Howie and colleagues introduced the concept of enablement, which represents patients' enablement, understanding of, and ability to cope with their health and illness. They developed the "The Patient Enablement Instrument" to measure patient competence based on the theory that if patients' competence increases, other important outcomes will improve. The Patient Enablement Instrument has since been translated into many languages and has generally demonstrated moderate to good validity and reliability. However, there are limitations to using the Patient Enablement Instrument as an outcome measure.

Inspired by the Patient Enablement Instrument, researchers from Denmark and Sweden developed the Patient Enablement Instrument for Back Pain , which could potentially be used as an outcome measure for interventions aimed at improving self-management in people seeking treatment for low back pain. In 2021, Nielsen et al. The validity and reliability of the scale was determined by and its use was recommended in the population experiencing low back pain. The aim of our study is to culturally adapt the Patient Enablement Instrument for Back Pain into Turkish and to examine its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain for at least 3 months

Exclusion Criteria:

* Having acute pain

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who have been experiencing low back pain for at least 3 months and agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-26 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Enablement Instrument for Back Pain | Baseline
  Each question is given a score between 0 and 10, allowing changes in the patient to be measured more sensitively. On a 0-10 numerical rating scale, 0 = "to a very low degree" and 10 = "to a very high degree". The maximum total score that can be obtained is 60, and higher scores indicate higher enablement.
Patient Enablement Instrument for Back Pain | After 1 week (retest)
  Each question is given a score between 0 and 10, allowing changes in the patient to be measured more sensitively. On a 0-10 numerical rating scale, 0 = "to a very low degree" and 10 = "to a very high degree". The maximum total score that can be obtained is 60, and higher scores indicate higher enablement.
The Brief Illness Perception Questionnaire | Baseline
  The scale consists of eight items. The eighth item on the scale questions the causal factors of the disease. The other 7 items in the scale have a Likert-type scoring scale from 0 to 10.
Fear-Avoidance Belief Questionnaire | Baseline
  It is a 16-item scale. It consists of 2 parts; The first part evaluates fear-avoidance attitudes related to physical activity, and the second part evaluates fear-avoidance attitudes related to work. Items with a 7-point Likert type receive a minimum of 0 points when the patient chooses the statement 'I completely disagree' and a maximum of 6 points when the patient chooses the statement 'I completely agree'.
Oswestry Low Back Pain Disability Questionnaire | Baseline
  It is a measurement method that evaluates daily life activities and consists of 10 questions. Questions include pain severity, personal care, weight lifting, walking, sitting, standing, sleep status, sexual and social life, and traveling. Each question consists of six items and is scored between 0-5.
Short Form 36 | Baseline
  The subscales of the scale are: physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems 31 (3 items), mental health (5 items), energy (4 items). item), pain (2 items) and general perception of health (5 items). Subscales evaluate health between 0 and 100, with 0 indicating the lowest quality of life and 100 indicating the highest quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Derived] Erol E, Arikan H. The patient enablement instrument for back pain turkish version, validity and reliability study. J Back Musculoskelet Rehabil. 2025 Sep;38(5):1044-1050. doi: 10.1177/10538127251322855. Epub 2025 Mar 25. PMID 40129386